CLINICAL TRIAL: NCT03831724
Title: Definition and Validation of Normative Data of EndoFLIP™ Measurements in Healthy Subjects ("RUBY Study")
Brief Title: Definition and Validation of Normative Data of EndoFLIP™ Measurements in Healthy Subjects
Acronym: RUBY
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Company decision to withdraw the study
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MDT18047
Record Dates: First submitted 2019-02-04; First posted 2019-02-06 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- EndoFLIP™ System (Experimental): Device interventions included in this arm: HRM, EGD including biopsies, EndoFLIP and Bravo
  Interventions: Device: EndoFLIP™ System with FLIP Topography Module

INTERVENTIONS:
Device: EndoFLIP™ System with FLIP Topography Module — The EndoFLIP system with the EF-322N catheter will be used. The EndoFLIP system is a tool that assesses esophageal, esophago-gastric junction (EGJ)/lower esophageal sphincter (LES), and pylorus function. It allows the measurement of LES and pylorus distensibility as well as esophageal contractile activity in response to distension. The system uses impedance planimetry to measure luminal cross-sectional area (CSA) along an axial plane during volume-controlled distention.

SUMMARY:
Multicenter, Prospective, Non-Randomized clinical trial to define and validate normative data of EGJ-distensibility measurements and contractile patterns in healthy subjects.

Asymptomatic subjects will be enrolled at up to 7 clinical sites in the United States.

Subjects who meet inclusion and no exclusion criteria and are deemed asymptomatic will be eligible for study enrollment.

The procedure visit/s will consist of the following procedures: High resolution manometry (HRM), esophagogastroduodenoscopy (EGD), endolumenal functional lumen imaging probe (EndoFLIP) and a Bravo procedure.

A post procedure follow-up phone call will be conducted within 5-9 days of completing all procedures.

HRM, EGD, and Bravo procedures are performed to evaluate subjects as normal in addition to being asymptomatic. Abnormal results in one or more of the procedures identifies the subject as unhealthy and the subject will be withdrawn from the study.

The expected duration of subject's participation in the study is up to 70 days (up to 30 days from screening to HRM, up to 30 days to complete EGD, EndoFLIP and Bravo, plus 5-9 days for follow up call).

Enrollment duration - up to 1 year

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female ages 18-75 years.
2. The subject has the ability to give informed consent.
3. The subject has the ability to undergo sedation, as assessed and determined by the treating physician or the anesthesiologist.
4. BMI range of 18-30 kg/m2.
5. Asymptomatic subjects as assessed by gastro-esophageal reflux disease questionnaire (GERDQ) negative score of less than 8 points (GERDQ <8) and brief esophageal dysphagia questionnaire (BEDQ) negative score of 0 points (BEDQ score=0), as assessed and determined by treating physician.

Exclusion Criteria:

1. Subject has known or suspected major gastrointestinal motility disorders including but not limited to major esophageal motility disorders, EGJ outflow obstruction and delayed gastric emptying.
2. Subject has dysphagia or any swallowing disorder.
3. Subject has an inability to tolerate nasal intubation.
4. Subject has a known or suspected bleeding diathesis.
5. Subject with known or suspected Gastroesophageal Reflux Disease (GERD), or subject has symptoms of GERD.
6. The subject has a known or suspected esophageal disease or disorder such as eosinophilic esophagitis (EOE), Barretts esophagus, severe esophagitis, upper GI bleeding or esophageal varices.
7. Subject is known or is suspected to suffer from an esophageal stricture or obstruction.
8. Subject has a hiatal hernia.
9. Subject with medical comorbidities such as diabetes, hypertension hyper/hypothyroidism, or chronic obstructive pulmonary disease (COPD)
10. Subject with a diagnosed autoimmune disease.
11. Subject who has undergone prior upper GI surgery or interventions such as esophageal myotomy, fundoplication, dilatation or stent.
12. Subject has a history of any malignancy.
13. Subject has a history of any seizure disorder.
14. Subject has a history of an eating disorder/s.
15. Subject has an active history of nicotine use, cannabis use or alcohol abuse (as defined by: greater than 14 drinks/week or 4 drinks/day for men, 7 drinks/week or 3 drinks/day for women. A standard drink is defined as 12 oz of beer, 5 oz of wine, or 1.5 oz of liquor). Subject has used any tobacco, nicotine or cannabis products in the last 6 months or has abused alcohol in the last 6 months.
16. Subject taking or prescribed or over-the-counter any acid suppressant medications (for example proton-pump inhibitors), any medication that treats reflux or heartburn symptoms (for example Tums and Maalox), any anticoagulant medications, any opiate medication or medication with known impact on GI motility.
17. Subject has any allergy or other contraindication to the device components or to study medication used prior and/or during the procedure.
18. Subject has a known sensitivity or allergy to nickel or other heavy metals.
19. Subject has any condition, which according to the investigators judgment, precludes compliance with study and/or device instructions.
20. Females who are pregnant or nursing at the time of screening and/or during the study period or are sexually active and of child bearing potential without medically acceptable methods of contraception.
21. Subject who has a cardiac pacemaker or implantable cardiac defibrillator.
22. Subject who has a general contraindication for upper endoscopy.
23. Subject who is currently participating in another clinical study (investigational drug or device).
24. Subject who is considered to be part of a vulnerable population (e.g. prisoners or those without sufficient mental capacity).
25. Medtronic employees.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Define and validate normative data of esophago-gastric junction -distensibility index (EGJ-DI) measurements at 60mL in healthy subjects | 70 days
  Median, 25% and 75% percentile for EGJ-DI measurements at 60mL balloon fill volume

SECONDARY OUTCOMES:
To define and validate normative data for an EGJ-DI at different balloon fill volumes within the same subject | 70 days
  Mean and median EGJ-DI at different balloon fill volumes of the same subject
To define and validate normative data for a maximum restrictive EGJ diameter at different balloon fill volumes within the same subject | 70 days
  Mean and median maximum restrictive EGJ diameter at different balloon fill volumes of the same subject
To define and validate normative data of a distal esophageal body diameter at different balloon fill volumes within the same subject | 70 days
  Mean and median distal esophageal body diameter at different balloon fill volumes of the same subject
To define and validate normative data of contractile patterns at different balloon fill volumes within the same subject | 70 days
  * Presence of Repetitive antegrade contractions (RACs) and number of antegrade contractions at different balloon fill volumes of the same subject
  * Presence of Repetitive Retrograde Contractions (RRCs) and number of retrograde contractions at different balloon fill volumes of the same subject

CONTACTS AND LOCATIONS:
Overall Officials: Rena Yadlapati, MD, Principal Investigator — University of Colorado, Denver

IPD SHARING:
Plan to Share IPD: No